CLINICAL TRIAL: NCT03522233
Title: Clinical Outcomes and Charges After Risk Stratification by Pediatric Appendicitis Risk Calculator (pARC) in Children With Appendix Ultrasounds at a Tertiary Care Pediatric Hospital
Brief Title: Pediatric Appendicitis Risk Calculator (pARC) in Children With Appendix Ultrasounds
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Children's Hospitals and Clinics of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 1708-113
Record Dates: First submitted 2018-04-18; First posted 2018-05-11 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-04

CONDITIONS: Appendicitis
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute appendicitis (AA) is the most common condition requiring emergency surgery in children. At a network of institutions nationwide, a tool called the pediatric appendicitis risk calculator (pARC)1 is being studied to assess patient's true risk of appendicitis and provide guidance for clinical management to ER physicians. Preliminary studies have found the pARC to be more accurate at predicting risk of appendicitis in children when compared to other scoring systems. The study objective is to assess acute care charges and clinical outcomes among children with an appendix ultrasound and a pARC score of less than < 25% risk.

DETAILED DESCRIPTION:
Background Acute appendicitis (AA) is the most common condition requiring emergency surgery in children. The potential for morbidity and mortality from perforation of the appendix necessitates prompt diagnosis.2 Acute appendicitis scoring systems such as pediatric appendicitis score (PAS) use elements of history, exam findings, and lab tests to identify patients at high risk of having acute appendicitis.3 Despite having limited use for this intent 4,5 these scores are often used to stratify patients by risk for continued observation, imaging or operative care. 6 While CT scans may have higher diagnostic yield, its use is not without risk. CT- related radiation exposure has been shown to increase cancer risk. There have been US first strategies published by the American College of Radiology7 and the American College of Emergency Physicians.8 However, nearly 50% of appendix US examinations are equivocal, which poses a dilemma for EM physicians and results in variation in clinical care.

Various strategies exist for the diagnostic approach to the patient after equivocal US with symptoms of AA. While select patients may be safely discharged based on clinical judgment,9 emergency providers often obtain CT or admit patients for clinical observation. In a study conducted by Garcia et al., they concluded that a protocol of US followed by CT in children with negative or equivocal US exam results in beneficial management as well as cost savings.10 In a study by Gregory et al., they concluded that a clinical decision rule followed by staged imaging was found to be the most cost-effective approach for diagnosis of AA in children.11 Bachur et al. integrated PAS score with US findings and concluded that patients with high risk (PAS 7-10) but negative US or low risk (PAS 0-3) benefit from serial exam or further work up. 12 The addition of US to the strategy reduced CT utilization.11 Standardized radiology reports have also been shown to reduce CT scans and admissions for observation.13 At a network of institutions nationwide a tool called the pediatric appendicitis risk calculator (pARC)1 is being studied to assess patient's true risk of appendicitis and provide guidance for clinical management to ER physicians. Preliminary studies have found the pARC to be more accurate at predicting risk of appendicitis in children when compared to PAS score.

The study objective is to assess acute care charges and clinical outcomes among children with appendix US and pARC < 25%. To the investigator's knowledge, this is the first study to do so in a tertiary care pediatric hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 5-18 years
* Patients who had an appendix ultrasound in one of our EDs

Exclusion Criteria:

* Outside appendix ultrasound or abdominal CT obtained
* Previous significant abdominal surgery (for example appendectomy, short gut, ileostomy, Hirschsprungs with pull through)
* No CBC obtained (i.e. cannot determine pARC)
* Developmental or cognitive delay that impedes communication
* If there is suspected abuse

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: We will collect data on all patients presenting to the emergency departments of Children's Minnesota between the ages of 5-18 years old who have a US of the appendix performed in the ED over 12 month period from September 23, 2017 to October 1, 2018.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2017-09-23 (Actual); Primary Completion 2018-10-01 (Estimated); Study Completion 2019-10-01 (Estimated)

PRIMARY OUTCOMES:
Rate of Equivocal Appendix Ultrasound | September 2017-October 2018
  To determine the rate of equivocal appendix US among children with pARC <25%.
Rate of Appendicitis | September 2017-October 2018
  To determine rate of appendicitis among children with pARC <25% who had an appendix ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Callie Becker, MD, Principal Investigator — Children's Minnesota
Locations (2):
- United States (2):
  - Children's Minnesota, Minneapolis, Minnesota
  - Children's Minnesota, Saint Paul, Minnesota

REFERENCES:
- [Background] Kharbanda AB, Vazquez-Benitez G, Ballard DW, Vinson DR, Chettipally UK, Kene MV, Dehmer SP, Bachur RG, Dayan PS, Kuppermann N, O'Connor PJ, Kharbanda EO. Development and Validation of a Novel Pediatric Appendicitis Risk Calculator (pARC). Pediatrics. 2018 Apr;141(4):e20172699. doi: 10.1542/peds.2017-2699. Epub 2018 Mar 13. PMID 29535251
- [Background] Pena BM, Taylor GA, Lund DP, Mandl KD. Effect of computed tomography on patient management and costs in children with suspected appendicitis. Pediatrics. 1999 Sep;104(3 Pt 1):440-6. doi: 10.1542/peds.104.3.440. PMID 10469767
- [Background] Samuel M. Pediatric appendicitis score. J Pediatr Surg. 2002 Jun;37(6):877-81. doi: 10.1053/jpsu.2002.32893. PMID 12037754
- [Background] Schneider C, Kharbanda A, Bachur R. Evaluating appendicitis scoring systems using a prospective pediatric cohort. Ann Emerg Med. 2007 Jun;49(6):778-84, 784.e1. doi: 10.1016/j.annemergmed.2006.12.016. Epub 2007 Mar 26. PMID 17383771
- [Background] Ebell MH, Shinholser J. What are the most clinically useful cutoffs for the Alvarado and Pediatric Appendicitis Scores? A systematic review. Ann Emerg Med. 2014 Oct;64(4):365-372.e2. doi: 10.1016/j.annemergmed.2014.02.025. Epub 2014 Apr 14. PMID 24731432
- [Background] Smith MP, Katz DS, Lalani T, Carucci LR, Cash BD, Kim DH, Piorkowski RJ, Small WC, Spottswood SE, Tulchinsky M, Yaghmai V, Yee J, Rosen MP. ACR Appropriateness Criteria(R) Right Lower Quadrant Pain--Suspected Appendicitis. Ultrasound Q. 2015 Jun;31(2):85-91. doi: 10.1097/RUQ.0000000000000118. PMID 25364964
- [Background] Howell JM, Eddy OL, Lukens TW, Thiessen ME, Weingart SD, Decker WW; American College of Emergency Physicians. Clinical policy: Critical issues in the evaluation and management of emergency department patients with suspected appendicitis. Ann Emerg Med. 2010 Jan;55(1):71-116. doi: 10.1016/j.annemergmed.2009.10.004. PMID 20116016
- [Background] Ross MJ, Liu H, Netherton SJ, Eccles R, Chen PW, Boag G, Morrison E, Thompson GC. Outcomes of children with suspected appendicitis and incompletely visualized appendix on ultrasound. Acad Emerg Med. 2014 May;21(5):538-42. doi: 10.1111/acem.12377. PMID 24842505
- [Background] Pena BM, Taylor GA, Fishman SJ, Mandl KD. Costs and effectiveness of ultrasonography and limited computed tomography for diagnosing appendicitis in children. Pediatrics. 2000 Oct;106(4):672-6. doi: 10.1542/peds.106.4.672. PMID 11015507
- [Background] Gregory S, Kuntz K, Sainfort F, Kharbanda A. Cost-Effectiveness of Integrating a Clinical Decision Rule and Staged Imaging Protocol for Diagnosis of Appendicitis. Value Health. 2016 Jan;19(1):28-35. doi: 10.1016/j.jval.2015.10.007. Epub 2015 Dec 2. PMID 26797233
- [Background] Bachur RG, Callahan MJ, Monuteaux MC, Rangel SJ. Integration of ultrasound findings and a clinical score in the diagnostic evaluation of pediatric appendicitis. J Pediatr. 2015 May;166(5):1134-9. doi: 10.1016/j.jpeds.2015.01.034. Epub 2015 Feb 21. PMID 25708690
- [Background] Partain KN, Patel AU, Travers C, Short HL, Braithwaite K, Loewen J, Heiss KF, Raval MV. Improving ultrasound for appendicitis through standardized reporting of secondary signs. J Pediatr Surg. 2017 Aug;52(8):1273-1279. doi: 10.1016/j.jpedsurg.2016.11.045. Epub 2016 Dec 5. PMID 27939802